CLINICAL TRIAL: NCT00663585
Title: Intensive Meditation and Migraines: Effects on Health and Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Madhav Goyal, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00016428; RR023266
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Daily Headache
Keywords: Migraine; Headache; Vipassana; Meditation; Intensive
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Structured Intervention Group
  Interventions: Behavioral: Vipassana Meditation
- 2.Comparison group (Active Comparator): Unstructured comparison group
  Interventions: Behavioral: Vipassana Meditation

INTERVENTIONS:
Behavioral: Vipassana Meditation — 12 day retreat where participants learn to meditate

SUMMARY:
Participants completing training in intensive meditation and continuing frequent practice for one year would experience reduced frequency, duration and severity of headaches along with improved awareness of the triggers of their symptoms, improved quality of life and mental health, improved heart rate variability, and reduced inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Daily Headache, defined as a headache at least 15 days of the month, of which at least 8 are migraines.

Exclusion Criteria:1.

* Severe depression, anxiety, panic attacks, psychosis or dementia that may interfere with ability to participate in a 10 day course
* Active alcoholism on screening or use of illicit drugs within the last 3 months
* Already completed a 10 day course
* Actively involved in another form of meditation over the past 6 months
* Women who are pregnant, planning pregnancy during trial period, or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
number of migraine days, number of headache days | 3,6,12 months

SECONDARY OUTCOMES:
severity of headaches | 3,6,12 months
quality of life | 3,6,12 months
Heart Rate Variability | 3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Goyal, MD, MPH, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Goyal M, Haythornthwaite JA, Jain S, Peterlin BL, Mehrotra M, Levine D, Rosenberg JD, Minges M, Seminowicz DA, Ford DE. Intensive Mindfulness Meditation Reduces Frequency and Burden of Migraine: An Unblinded Single-Arm Trial. Mindfulness (N Y). 2023 Feb;14(2):406-417. doi: 10.1007/s12671-023-02073-z. Epub 2023 Jan 24. PMID 38282695